CLINICAL TRIAL: NCT00001604
Title: Genetic Studies of Stuttering
Brief Title: Genetic Linkage Studies of Stuttering
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970057; 97-DC-0057
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Stuttering
Keywords: DNA Samples; Stuttering; DNA Testing; Statistical Analysis; Genetic Analysis; Natural History
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subjects with a family history of stuttering

SUMMARY:
Stuttering is an abnormality in speech that affects the rhythm of speech. People who stutter know what they wish to say, but at the time are unable to say it because of involuntary repetition, unnecessary lengthening (prolongation), or early stopping (cessation). Stuttering is characterized by repetitions or prolongation of the first syllable, or silent prolongations, sometimes known as blocks.

Researcher intend on studying the genetic basis for stuttering. The goal of the study is to find the genes that help cause stuttering and determine regions of the human genetic make-up (genome) that are linked to stuttering.. To do this researchers will study the patterns of inheritance in families who have had members who stutter.

The study has two objectives.

The first objective is to develop a large collection of DNA samples from individuals in stuttering families, that will include both members that stutter and who do not stutter.

The second objective of the study will be to find out the basic combination of genes (genotype) making up all of the participants DNA. Once this is completed researchers hope to map out and find areas or regions of DNA that are linked to stuttering.

Genetic linkage is the initial step in positional cloning, and the cloning of genes which predispose individuals to stuttering is a long term goal of this research study.<TAB>

DETAILED DESCRIPTION:
A primary goal of this study is to ascertain regions of the human genome which show genetic linkage to stuttering. Genetic linkage will be determined by first obtaining genomic DNA from both affected and unaffected adults and children from families containing pairs of individuals who stutter as adults. Individuals who stutter from genetically isolated populations will also be sampled. Phenotype will be assigned by a speech-language pathologist, and DNA samples will be obtained from affected and unaffected family members from 2 cc. of saliva or from 20 cc. of blood. These DNA samples will then be genotyped using markers distributed across the human genome. The genotypic information analyzed to determine which markers or variants show linkage to stuttering. The initial goal of this study is to identify specific genetic variants, which predispose individuals to stuttering. No genetic information will be provided back to participants. A secondary goal of the study will be to perform broad clinical evaluations of the individuals found to have mutations that cause stuttering. These will take place at the NIH Clinical Center and will include standard procedures including history and physical, neurological exam, audiological exam, ophthalmologic exam, electromyographic (EMG) exam, electroencephalography (EEG), X-rays, speech evaluation, and brain imaging including MRI and fMRI.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals age 8 and older.
* Individuals age 6-8 with a family history of persistent stuttering
* Have stuttering that persists for a period of 6 months or more or are a family member of that person
* For the Phase 2 imaging studies, we will be enrolling up to 25 healthy volunteers to be controls

EXCLUSION CRITERIA:

* Stuttering only as a young child (before age 5) with no other family members who stutter
* Inability to provide informed consent or have a parent/guardian to provide consent
* Development of stuttering following trauma to the central nervous system.
* Chronic medical conditions that prevent informed consent or clear evaluation of stuttering, including stroke, dementia, and degenerative neurological disease.
* Inability to travel to the NIH Clinical Center for Phase 2

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected primarily on the basis of family history of stuttering. Certain populations, such as those in Pakistan present increased power to detect genetic influences on stuttering, and such populations will be preferentially enrolled where possible and appropriate. No one will be excluded on the basis of gender or ethnic/racial background.
Sampling Method: Non-Probability Sample
Enrollment: 3044 (Actual)
Dates: Start 2003-07-22 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
To identify genetic mutations or variants that predispose humans to stuttering. | ongoing
  Our primary outcome measures are the observation or exclusion of genetic linkage to stuttering at a discreet locus or genetic association with stuttering with a specific genetic variant.

SECONDARY OUTCOMES:
Perform clinical and physical evaluations on those individuals who stutter and possess these genetic variants | ongoing
  disorders in study subjects carrying genetic variants shown to be associated with stuttering in the primary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Levy, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (3):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- National Rehabilitation Center for Persons with Disabilities Hospital, Saitama, Japan
- NCEMB - University of Punjab, Lahore, Pakistan

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-DC-0057.html